CLINICAL TRIAL: NCT00877539
Title: A Randomized, Double-Blind, Double-Dummy, Placebo Controlled, 3-Way Crossover Study To Determine The Effects Of Inhaled Doses Of PF-03526299 On Allergen-Induced Airway Responses In Mild Asthmatic Subjects.
Brief Title: A Study To Assess The Effect Of PF-03526299 On Lung Function Following An Allergen Challenge In Asthmatic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A9291002
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Asthma
Keywords: Asthma Allergen Challenge
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-03526299 (Experimental)
  Interventions: Drug: PF-03526299
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Fluticasone propionate (Active Comparator)
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: PF-03526299 — Inhaled, two doses 4 hours apart
  Arms: PF-03526299
Drug: Placebo — Inhaled, two doses 4 hours apart
  Arms: Placebo
Drug: Fluticasone propionate — Inhaled
  Arms: Fluticasone propionate

SUMMARY:
PF-03526299, a novel anti-inflammatory agent should attenuate the effect of a bronchial allergen challenge on lung function and hence provide proof of mechanism for this agent.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-60 years
* Mild asthma
* Atopic to allergens

Exclusion Criteria:

* Unstable asthma
* Smokers or recent ex-smokers
* Recent allergen challenge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Spirometry pre- and post- bronchial allergen challenge | 2 months

SECONDARY OUTCOMES:
Laboratory safety tests | 2 months
12-lead ECGs | 2 months
Adverse Event reporting | 2 months
Blood samples for pharmacokinetic measurement | 2 months
Sputum for pharmacodynamic measurement | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United Kingdom (2):
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9291002&StudyName=A%20Study%20To%20Assess%20The%20Effect%20Of%20PF-03526299%20On%20Lung%20Function%20Following%20An%20Allergen%20Challenge%20In%20Asthmatic%20Subjects